CLINICAL TRIAL: NCT03420326
Title: The Relationship Between Atrial Fibrillation and Frailty in Community-Dwelling
Brief Title: The Relationship Between Atrial Fibrillation and Frailty in Community-Dwelling Elderly
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201711083RIND
Record Dates: First submitted 2018-01-25; First posted 2018-02-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Frail Elderly Syndrome
Keywords: Atrial Fibrillation; Frailty status; Body composition; Sarcopenia
MeSH Terms: conditions — Atrial Fibrillation; Sarcopenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atria fibrillation (AF) group: 1. Detection of AF during 30 seconds ECG assessment
  2. Once diagnosed with atrial fibrillation before
  3. Undergo the frailty status assessment
  Interventions: Behavioral: Frailty status assessment
- Non-AF group: 1. No detection of AF during 30 seconds ECG assessment
  2. Undergo the frailty status assessment
  Interventions: Behavioral: Frailty status assessment

INTERVENTIONS:
Behavioral: Frailty status assessment — The Edmonton frail scale and Frailty criteria by Dr. Fried would be used to assess participants frailty status

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmias in clinical practice. Research investigating hospitalized patients have indicated there are deleterious effects of AF on patients besides the disease burden itself, including longer stay days for hospitalization, higher rates of frailty and increasing mortality rate after discharged in six months. In the community-dwelling research also found that elderly with AF have lower cognitive function, physical functional tests score and slower walking speed compared with the health ones. However, there is limited articles investigating the impact of AF on community-dwelling elderly, and the relationship between AF and frailty is also lack of discussion. According to the aged society and increasing prevalence of AF, the relationship between AF and frailty in community-dwelling elderly is warranting investigated.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years old

Exclusion Criteria:

diagnosed with the following disease

1. Cardiovascular diseases: myocardial infarction, peripheral vascular diseases, aortic plaque
2. Cerebrovascular disease: stroke, transient ischemic attack, emboli
3. Heart failure
4. Participants who cannot finish the trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: National Taiwan University Hospital Communities in Taipei city
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Frailty status | The frail status assessment would take about 10 minutes
  Edmonton frail scale and Frailty criteria by Dr. Fried would be used to evaluate the frail status of the participants

SECONDARY OUTCOMES:
Body composition | The body composition test would take about 10 minutes
  Maltron BioScan BF-920, Essex, UK would be used to assess participants' body composition

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, Study Chair — College of medicine, National Taiwan University
Locations (1):
- Ming-Ting Yang, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided